CLINICAL TRIAL: NCT04640636
Title: IM Ketamine vs Midazolam for Suicidal ER Patients
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Grunebaum, MD, Research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8070-76595; R01MH125155-01 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Depression, Unipolar; Depression, Bipolar; Suicidal Ideation
Keywords: depression; suicidality; clinical trial; ketamine; midazolam
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Suicidal Ideation; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Ketamine hydrochloride 0.5 mg/kg IM single injection
  Interventions: Drug: Ketamine hydrochloride injection
- midazolam (Active Comparator): Midazolam 0.06 mg/kg IM single injection
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Ketamine hydrochloride injection — single IM injection of ketamine hydrochloride 0.5 mg/kg
  Arms: Ketamine
Drug: Midazolam injection — single IM injection of midazolam 0.06 mg/kg
  Arms: midazolam

SUMMARY:
Rising US suicide rates and the increased risk of suicide among persons who visit an emergency department (ED) for suicidality make the ED an important site for interventions to prevent suicide. There is no approved treatment for rapid relief of suicidal thoughts although clinical trials, including ours, show relief of suicidal thoughts within hours of treatment with inexpensive, generic, sub-anesthetic ketamine. We propose a clinical trial of intramuscular ketamine in depressed ED patients with high-risk suicidality, which if successful would support a novel, easy-to-use, scalable intervention for busy emergency clinicians to implement.

NOTE: The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June, 2023.

The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.

Non-HHS Studies: The IO in concurrence with the IRB paused human subjects research on June 12, 2023. Therefore, the NYSPI site is not enrolling at this time.

DETAILED DESCRIPTION:
Rising US suicide rates and the increased risk of suicide among persons who visit an emergency department (ED) for suicidality make the ED an important site for interventions to prevent suicide. Clinical trials, including ours, show relief of suicidal thoughts within hours of treatment with inexpensive, generic, subanesthetic ketamine. We have received NIMH R01 funding to conduct a clinical trial of intramuscular (IM) ketamine in unipolar or bipolar depressed adults who present to the CUIMC psychiatric ED with suicidality severe enough to require inpatient hospitalization as judged by ED clinical staff. Clinical staff will ask potentially eligible patients if they would like to learn more about the study, and if so, a research assistant (RA) will describe the study to the patient and perform a basic eligibility screen. Key exclusions are unstable medical problems, substance abuse, psychosis, and further detail is provided in the Inclusion/Exclusion criteria. Participants (N=90) who enroll will undergo baseline clinical ratings, brief cognitive testing, and then be randomized, double-blind, in a 2:1 ratio to a single IM injection of ketamine (n=60) or midazolam comparator (n=30). Vital signs and clinical state will be monitored until injection effects subside (approximately 2 hrs). Blood samples will be drawn at 60 minutes and 90 minutes postinjection to assay ketamine level and a genetic sample will be stored. All participants will then be admitted to the 9GN inpatient unit for standard clinical treatment with periodic research follow-up ratings through 4 weeks post-discharge from hospital. Ongoing outpatient treatment will be arranged by the inpatient clinical team. Positive results from this trial would support a novel, easy-to-use, inexpensive, and scalable intervention for busy emergency clinicians to implement.

ELIGIBILITY:
Inclusion Criteria:

* DSM5 unipolar or bipolar (I, II, or Unspecified) major depressive episode
* Presenting to emergency department and assessed by psychiatrist staff as needing inpatient treatment due to suicidality
* Participant agrees to voluntary inpatient psychiatric admission
* Beck Scale for Suicidal Ideation score of 4 or higher

Exclusion Criteria:

* Substance use disorder in past 2 weeks
* Current psychosis or mania
* Intellectual disability
* Inadequate understanding of English and/or lack of capacity for informed consent
* Pregnancy or lactation
* Medical contraindication to ketamine or midazolam
* Unstable medical or neurological illness such as uncontrolled hypertension, significant cardiac arrhythmia, unstable cerebrovascular disease. Chronic, stable medical conditions such as controlled hypertension or diabetes will not be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicidal Ideation (SSI) | 24 hours post-treatment
  Beck Scale for Suicidal Ideation clinician-rated version

SECONDARY OUTCOMES:
Systematic Assessment for Treatment Emergent Events (SAFTEE) | 24 hours post-treatment
  Frequency of adverse events at 24 hours post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grunebaum, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University Irving Medical Center
Locations (1):
- Comprehensive Psychiatric Emergency Department of Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All associated research findings published or provided to NIH, will be made readily available for research purposes to qualified individuals within the scientific community. All data will be made anonymous and available after written requests for data are submitted by such qualified individuals to the PI.
Supporting Information: Study Protocol, SAP, ICF